CLINICAL TRIAL: NCT01764412
Title: Study of Serum Hepcidin Rate Variations During Menstrual Cycle
Acronym: HEPMEN
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A01122-41
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Women
Keywords: Healthy women; Menstrual cycle; Hepcidin; Seric iron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hepcidin Serum iron Transfferin saturation Serum transfferin Serum ferritin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy women: Non interventional

SUMMARY:
Hepcidin is the major hormone regulating Iron Metabolism. In a normal organism decrease iron stock causes a decrease in hepcidin synthesis thus promoting intestinal absorption of iron.

The interpretation of hepcidin dosage results requires to know the physiological variations of this hormone.

This study investigate whether there are significant variations in the values of serum hepcidin rates during the menstrual cycle in order to make recommendations on the practical dosage determination of hepcidin in premenopausal women.

DETAILED DESCRIPTION:
Hepcidin is the major hormone regulating Iron Metabolism. Synthesized primarily by hepatocytes, it interacts with the cellular iron exporter ferroportin, causing its internalization and preventing the release of iron from enterocytes and macrophages.

In a normal organism decrease iron stock causes a decrease in hepcidin synthesis thus promoting intestinal absorption of iron.

Since valid methods for the determination of hepcidin serum rate are available, this dosage is increasingly used to diagnosis iron metabolism pathologies, in particular iron overload. The interpretation of hepcidin dosage results requires to know physiological variations of this hormone.

Several works have shown that hepcidin varies according to a circadian cycle, that its values differ by sex and, in women, by age. As far as the investigators know, no study has focused on possible variations in serum hepcidin rates values during menstrual cycle in women. Yet this question seems relevant since it has been shown that during the menstrual cycle blood loss can cause significant iron and hemoglobin variations, which can significantly modulate the synthesis of hepcidin.

This study investigate whether there are significant variations in the values of serum hepcidin rates during the menstrual cycle in order to make recommendations on the practical dosage determination of hepcidin in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged over 18 and under 45 years,
* Having given free and informed written consent,
* Having regular cycles (defined by a constant interval between periods of 28 to 30 days),
* Having periods for a duration of 4 + / - 1 days
* Not using contraception or using oral oestroprogestative contraception.

Exclusion Criteria:

* Contraceptive IUD
* Metrorrhagia
* Pregnancy,
* BMI under 18 kg / m² and above 30 kg / m²,
* Presence of at least one of the following abnormalities in serum iron balance : Hemoglobin <11.5 g / dl, transferrin saturation under 15% or greater than 50%, serum ferritin under 15μg / l or greater than 150 µg / l
* Active smoking or quit within the last 6 months
* Drinking more than 20 g of alcohol per day ,
* Iron supplementation or blood transfusion within 12 months before inclusion
* Blood donation within 3 months before inclusion,
* Stay in altitude> 1500 m in the previous month before inclusion
* Chronic inflammatory disease,
* Incapable people over 18 (judicial protection, guardianship) and persons deprived of their liberty.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Serum hepcidin rates variations during the menstrual cycle | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26

SECONDARY OUTCOMES:
Seric iron | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26
transferrin saturation | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26
serum transferrin | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26
serum ferritin | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26
hepcidin / ferritin rate | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26
hepcidin / transferrin saturation rate | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26
hepcidin / serum iron rate | During the menstrual cycle (see description)
  Time frame : depending on the calendar day of D1 as the following calendars (D1: first day after periods beginning)
  * D1 occurring on Monday : D1, D3, D4, D8, D15, D26
  * D1 occurring on Tuesday : D1, D2, D4, D7, D11, D28
  * D1 occurring on Wednesday : D1, D2, D6, D7, D13, D28
  * D1 occurring on Thursday : D1, D2, D5, D6, D13, D28
  * D1 occurring on Friday : D1, D4, D5, D6, D11, D27
  * D1 occurring on Saturday : D3, D4, D5, D12, D20, D27
  * D1 occurring on Sunday : D3, D4, D5, D12, D19, D26

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice lainé, MD, Principal Investigator — CHU de Rennes - CIC INSERM 0203
Locations (4):
- France (4):
  - CHU Rennes, Rennes, Brittany Region
  - Chu Brest, Brest
  - CHU Nantes, Nantes
  - Chru Tours, Tours